CLINICAL TRIAL: NCT04968964
Title: TK IMPACT: Treatment Monitoring of Patients Receiving CDK 4/6 Inhibitors for Hormone Receptor (HR) Positive, HER2 Negative Metastatic Breast Cancer (MBC) With or Without the Addition of DiviTum® Serum Thymidine Kinase 1 (TK1) Activity Testing: Physician Decision Impact Study
Brief Title: Treatment Monitoring of Patients Receiving CDK 4/6 Inhibitors for Hormone Receptor (HR) Positive, HER2 Negative Metastatic Breast Cancer (MBC) With or Without the Addition of DiviTum® Serum Thymidine Kinase 1 (TK1) Activity Testing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Biovica (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202107015
Record Dates: First submitted 2021-07-08; First posted 2021-07-20 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer; Cancer of the Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Cohort 1: Scheduled to receive first line therapy (Experimental): * Scheduled to receive 1st line therapy with endocrine therapy + any FDA-approved CDK 4/6 inhibitor
  * Serum samples (analyzed using DiviTum® TKa) at Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 20, Week 24 and every 12 weeks thereafter until disease progression or 36 months. Treating physician will evaluate the patient & review any updated results of the institutional standard of care monitoring tests. Following receipt of DiviTum® TKa value, the treating physician will review the preceding locked Study Care Plan and record any changes
  Interventions: Device: DiviTum® TKa assay
- Cohort 2: Currently receiving first line therapy (Experimental): * 1st line therapy with endocrine therapy + any FDA-approved CDK 4/6 inhibitor for ≤ 24 months with stable disease
  * Serum samples (analyzed using DiviTum® TKa) at Baseline, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 20, Week 24 and every 12 weeks thereafter until disease progression or 36 months. Treating physician will evaluate the patient & review any updated results of the institutional standard of care monitoring tests. Following receipt of DiviTum® TKa value, the treating physician will review the preceding locked Study Care Plan and record any changes
  Interventions: Device: DiviTum® TKa assay
- Medical Oncologists (Experimental): -Will be completing the Study Care Forms at Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 and every 12 weeks thereafter until disease progression or 36 months.
  Interventions: Other: Study Care Plans

INTERVENTIONS:
Device: DiviTum® TKa assay — -Determines serum enzymatic activity of TK1
  Arms: Cohort 1: Scheduled to receive first line therapy; Cohort 2: Currently receiving first line therapy
Other: Study Care Plans — -Study Care Plans will be completed prior to and post release of serum DiviTum® TKa value
  Arms: Medical Oncologists

SUMMARY:
Historically, serial testing of patients with metastatic breast cancer has included a combination of physical exam, symptom evaluation, laboratory testing, and imaging. Circulating tumor biomarkers are sometimes also incorporated. Frequent testing with numerous diagnostics at each time point is a significant burden to patients and to healthcare systems.

The DiviTum® TKa assay measures TK1 activity. Numerous studies have illustrated the prognostic nature of plasma or serum TK1 activity level in metastatic cancer. The investigators hypothesize that the incorporation of data from DiviTum® TKa measurement into the treatment monitoring schema will be associated with physician desire to change the near-term usage and/or timing of other routine restaging tests, including either standard tumor imaging or tumor marker testing. Given the relatively low rate of disease progression in this first-line population, it is expected that most of this change will be an intended reduction in scheduling of routine treatment surveillance testing with increase in intervals of subsequent tumor restaging imaging by at least 4 weeks. Secondarily, the consequences of rescheduling of routine surveillance testing may ultimately result in an absolute reduction in the number of some tests used during the time period examined.

ELIGIBILITY:
Inclusion Criteria - Patients:

* Diagnosis of metastatic or advanced resectable invasive breast cancer that is hormone receptor-positive (HR+) and HER2-negative. Tumor assessment by radiographic imaging will be performed within 4 weeks of baseline study visit.
* Cohort 1 only: Scheduled to initiate standard of care first-line combination therapy with any FDA-approved endocrine therapy plus any FDA-approved CDK 4/6 inhibitor (palbociclib, ribociclib, or abemaciclib) for the stated diagnosis at the time of study enrollment. Type of endocrine therapy and CDK 4/6 inhibitor will be documented. Patients may also be eligible if:

  * Patients were treated with and progressed on prior endocrine therapy monotherapy in the metastatic setting, OR
  * Patients initiated endocrine therapy alone with ultimate intention to add CDK 4/6 inhibitor therapy, OR
  * Patients recurred on adjuvant endocrine therapy monotherapy and are scheduled to receive next line endocrine therapy combined with CDK 4/6 inhibitor. Patients may have also received CDK 4/6 inhibitor therapy in the adjuvant setting provided therapy completion occurred greater than 12 months prior to study enrollment.
* Cohort 2 only: Currently receiving first-line combination therapy with any FDA-approved endocrine therapy plus any FDA-approved CDK 4/6 inhibitor (palbociclib, ribociclib, or abemaciclib). Changes in endocrine therapy or CDK 4/6 inhibitor agent during first-line combination therapy are permitted as long as change was not performed due to progressive disease. CDK 4/6 inhibitor must have been initiated within 24 months of study enrollment, and patient must have at least stable disease (no progression) on such therapy for a minimum of 12 weeks prior to enrollment as determined by radiographic studies as deemed appropriate by the treating physician. Type of endocrine therapy and CDK 4/6 inhibitor will be documented. Patients may also be eligible if they are receiving next line endocrine therapy plus CDK 4/6 inhibitor therapy following:

  * Progression on prior endocrine therapy monotherapy in the metastatic setting, OR
  * Recurrence on adjuvant endocrine therapy monotherapy. Patients may have also received CDK 4/6 inhibitor therapy in the adjuvant setting provided therapy completion occurred greater than 12 months prior to study enrollment.
* Any prior therapy for early stage breast cancer is allowed, including endocrine therapy and chemotherapy.
* At least 18 years of age.
* Life expectancy > 6 months.
* Post-menopausal status, defined as one of the following:

  * Age ≥ 60 years
  * Age < 60 with intact uterus and amenorrhea for 12 consecutive months or more
  * Status post bilateral oophorectomy, total hysterectomy
  * Pre- or peri-menopausal with suppressed ovarian function by use of GnRH agonist/antagonist or surgical bilateral oophorectomy
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).
* Currently being treated at Siteman Cancer Center by a medical oncologist participating in this trial.

Exclusion Criteria - Patients:

* Receipt of any prior cytotoxic chemotherapy line for metastatic disease. There will be no limited to chemotherapy use in the neoadjuvant or adjuvant setting.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the protocol assessments or analyses are eligible for this trial as determined by treating physician and with agreement by Principal Investigator
* Concurrent participation in any investigational therapeutic trial for treatment of metastatic breast cancer.

Eligibility Criteria - Physicians:

* Medical Oncologist at Siteman Cancer Center
* Treating patients with metastatic or advanced unresectable invasive breast cancer
* Willing to complete Study Care Plans on a serial basis during participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Any physician-reported intended change in imaging testing interval identified on the study care plan post receipt of DiviTUM® TKa value | Within the first 48-week period of study participation

SECONDARY OUTCOMES:
Concordance rate between progression status on the first on-study imaging and progression status based on DiviTum® TKa values | At 12 weeks
Concordance rate between progression status on the first on-study imaging and progression status based on DiviTum® TKa values | At 12 weeks and 24 weeks
Number of surveillance imaging tests intended to be used and actually used, in total and by modality | Over the entire study period (estimated to be 36 months)
Longitudinal changes in DiviTum® TKa value dynamics | Over the entire study period (estimated to be 36 months)
  The TK trajectory of a patients will be plot against time for temporal pattern and the trajectories will be modeled via linear or non-linear mixed effects mode as appropriate. If linear mixed effects model, the longitudinal rate of change will be estimated with 95% CI to indicate growth rate of TK. If non-linear, the regression coefficients of time or time relevant terms will be estimated with 95% CI
Cohort 1 only: DiviTum® TKa level | At 2 weeks post CDK 4/6 inhibitor therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Nusayba Bagegni, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu